CLINICAL TRIAL: NCT07255963
Title: A Prospective Study of Pirtobrutinib, Lisaftoclax, and Rituximab in the Treatment of Relapsed or Refractory Diffuse Large B-Cell Lymphoma (R/R DLBCL)
Brief Title: Pirtobrutinib, Lisaftoclax, and Rituximab in the Treatment of R/R DLBCL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025807
Record Dates: First submitted 2025-09-26; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: DLBCL - Diffuse Large B Cell Lymphoma
Keywords: pirtobrutinib; Lisaftoclax; DLBCL
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating | interventions — pirtobrutinib; Lisaftoclax; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pirtobrutinib, Lisaftoclax, and Rituximab (Experimental): R/R DLBCL patients will receive PVR for a total of 2 treatment cycles (28 days per cycle) in the induction treatment. Patients with CR/PR after two cycles recieve consolidation therapy : ASCT or CAR-T or PVR (R for 6 cycles, PV continued until disease progression or intolerable adverse reactions) or radiotherapy.The patient will be followed up for two years.
  Interventions: Drug: Pirtobrutinib; Drug: Lisaftoclax; Drug: Rituximab

INTERVENTIONS:
Drug: Pirtobrutinib — 200mg qd po
Drug: Lisaftoclax — cycle 1: 200mg qd d1-7; 400mg qd d8-d28；Cycle 2: 400mg qd d1-d28 po
Drug: Rituximab — 375mg/m2 d1 intravenous drip

SUMMARY:
This study aims to evaluate the efficacy of combining pirtobrutinib, lisaftoclax, and rituximab (PVR) in patients with relapsed or refractory diffuse large B-cell lymphoma (DLBCL) who have received at least one prior line of systemic therapy and to explore a more effective treatment strategy for this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old.
2. Capable of understanding and voluntarily signing written informed consent.
3. ECOG performance 0 ~ 3.
4. Anticipated survival ≥3 months
5. Histologically or cytologically confirmed DLBCL.
6. PET-CT-defined measurable disease with a short axis diameter of ≥1.5 cm.
7. Have received at least one prior line of systemic therapy for DLBCL.
8. Resolution of any prior treatment-related non-hematologic toxicities to Grade ≤1 or baseline.
9. Adequate Bone Marrow and Organ Function, defined as:

   Bone Marrow Function: ANC≥1.5 × 10⁹/L, Platelets ≥80 × 10⁹/L, Hemoglobin ≥80 g/L Hepatic Function: Total bilirubin ≤1.5 × ULN (≤3.0 × ULN if liver metastases present); AST/SGOT and ALT/SGPT ≤2.5 × ULN (≤5.0 × ULN if liver metastases present) Coagulation: INR and aPTT≤1.5 × ULN Renal Function: Serum creatinine ≤1.5 × ULN or estimated creatinine clearance (CrCl) ≥60 mL/min;
10. Subjects with childbearing or childbearing potential must be willing to practice birth control from the date of registration in this study to the follow-up period of the study.
11. Able to swallow tablets/capsules without difficulty.
12. Adhere to scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Prior treatment failure or resistance to pirtobrutinib or BCL2 inhibitors.
2. Prior Anticancer Therapy:Chemotherapy, radiotherapy, immunotherapy, or antibody-based anticancer therapy within the specified washout period.Traditional Chinese herbal medicine with antitumor indications.Small-molecule targeted therapy within 2 weeks before study treatment initiation. ADCs or cytotoxic therapy within 10 weeks before study treatment initiation.
3. Participation in another investigational drug study within 4 weeks prior to the first dose of study treatment.
4. Systemic corticosteroid therapy (>5 days within 14 days prior to treatment) at doses exceeding >10 mg/day dexamethasone (or equivalent) for CNS disease control.
5. Requiring ongoing anticancer therapy.
6. Uncontrolled or Severe Cardiovascular Disease,
7. Active infection requiring IV antibiotics or systemic antimicrobial therapy.
8. Active HBV/HCV:Exceptions. Inactive HBsAg carriers, HBV patients with sustained viral suppression (HBV-DNA < LLOD),HCV-cured patients are allowed.
9. Clinically significant abnormalities affecting drug absorption or prior total gastrectomy/gastric banding.
10. History of hemorrhagic diathesis or requirement for long-term oral anticoagulation.
11. Prior allogeneic hematopoietic stem cell transplantation (HSCT) or planned allogeneic HSCT.
12. Women who are pregnant or breastfeeding.
13. Known allergy to the study drug or its excipients.
14. Active psychiatric illness or history of alcohol/drug abuse .
15. Any uncontrolled illness, organ dysfunction, or medical condition that, in the investigator's judgment, jeopardizes patient safety or adherence to study procedures.
16. Other conditions deemed inappropriate for study participation by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | At the end of 2 cycles of PVR regimen (each cycle is 28 days)
  The rate of patients who achieved CR or PR after 2 cycles of PVR regimen

SECONDARY OUTCOMES:
Complete response rate(CRR) | At the end of 2 cycles of PVR regimen (each cycle is 28 days)
  The rate of patients who achieved CR after 2 cycles of PVR regimen
Adverse Events | During induction treatment
  The safety during induction treatment

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou Z, Zhang L, Wang X, Li X, Li L, Fu X, Zhang X, Li Z, Sun Z, Zhang M. Ibrutinib combined with venetoclax for the treatment of relapsed/refractory diffuse large B cell lymphoma. Ann Hematol. 2021 Jun;100(6):1509-1516. doi: 10.1007/s00277-021-04535-7. Epub 2021 Apr 26. PMID 33900450
- [Background] Roeker LE, Woyach JA, Cheah CY, Coombs CC, Shah NN, Wierda WG, Patel MR, Lamanna N, Tsai DE, Nair B, Wang C, Zhao X, Liu D, Radtke D, Chapman S, Marella N, McNeely SC, Brown JR. Fixed-duration pirtobrutinib plus venetoclax with or without rituximab in relapsed/refractory CLL: the phase 1b BRUIN trial. Blood. 2024 Sep 26;144(13):1374-1386. doi: 10.1182/blood.2024024510. PMID 38861666